CLINICAL TRIAL: NCT03334747
Title: A Phase 2, Multi-center, Randomized, Open-label, Dose-escalation Study to Determine Safety of Single (QD) and Multiple (3 QD) Doses of KAE609, Given to Adults With Uncomplicated Plasmodium Falciparum Malaria.
Brief Title: Safety of KAE609 in Adults With Uncomplicated Plasmodium Falciparum Malaria.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKAE609A2202; 207813/Z/17/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2017-10-27; First posted 2017-11-07 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Malaria
Keywords: uncomplicated Plasmodium falciparum Malaria.
MeSH Terms: conditions — Malaria | interventions — NITD 609; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: Patients were randomized to KAE609 and Coartem in parallel treatment arms. Increasing doses of KAE609 (single dose and multiple dose) were evaluated in dose escalated manner in sequential cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Treatment arm 1: KAE609 10 mg Single Dose (SD) (Experimental): KAE609 10 mg once daily (QD) for 1 day
  Interventions: Drug: KAE609
- Treatment arm 2:KAE609 25 mg SD (Experimental): KAE609 25 mg once daily (QD) for 1 day
  Interventions: Drug: KAE609
- Treatment arm 3:KAE609 10 mg 3 Days (Experimental): KAE609 10 mg (QD) for 3 days
  Interventions: Drug: KAE609
- Treatment arm 4:KAE609 50 mg SD (Experimental): KAE609 50 mg once daily (QD) for 1 day
  Interventions: Drug: KAE609
- Treatment arm 5:KAE609 25 mg 3 Days (Experimental): KAE609 25 mg once daily (QD) for 3 days
  Interventions: Drug: KAE609
- Treatment arm 6:KAE609 75 mg SD (Experimental): KAE609 75 mg once daily (QD) for 1 day
  Interventions: Drug: KAE609
- Treatment arm 7:KAE609 50 mg 3 Days (Experimental): KAE609 50 mg once daily (QD) for 3 days
  Interventions: Drug: KAE609
- Treatment arm 8: KAE609 150 mg SD (Experimental): KAE609 150 mg once daily (QD) for 1 day
  Interventions: Drug: KAE609
- Treatment arm 9: Coartem Control (Active Comparator): Coartem® control
  Interventions: Drug: Coartem

INTERVENTIONS:
Drug: KAE609 — Exploration of different doses of KAE609 to establish safety profile.
  Other Names: Cipargamin
  Arms: Treatment arm 1: KAE609 10 mg Single Dose (SD); Treatment arm 2:KAE609 25 mg SD; Treatment arm 3:KAE609 10 mg 3 Days; Treatment arm 4:KAE609 50 mg SD; Treatment arm 5:KAE609 25 mg 3 Days; Treatment arm 6:KAE609 75 mg SD; Treatment arm 7:KAE609 50 mg 3 Days; Treatment arm 8: KAE609 150 mg SD
Drug: Coartem — Control Arm
  Other Names: Artemether Lumefantrine
  Arms: Treatment arm 9: Coartem Control

SUMMARY:
KAE609 will be evaluated primarily for hepatic safety of single and multiple doses in sequential cohorts with increasing doses.This study aims to determine the maximum safe dose of the investigational drug KAE609 in malaria patients.

ELIGIBILITY:
KEY Inclusion Criteria:

1. Male and female patients ≥ 18 years with a body weight ≥ 45 kg.
2. Microscopic confirmation of acute uncomplicated P. falciparum using by Giemsa-stained thick film.
3. P. falciparum parasitaemia of 500 to 50 000 parasites/µL.
4. Axillary temperature ≥ 37.5ºC or oral/tympanic/rectal temperature ≥ 38.0ºC; or history of fever during the previous 24 hours.
5. Written informed consent must be obtained before any study assessment is performed. If the patient is unable to write, then a witnessed consent according to local ethical standards is permitted.

KEY Exclusion Criteria:

1. Mixed Plasmodium infections.
2. Signs and symptoms of severe malaria according to World Health Organization (WHO) 2016 criteria (WHO 2016).
3. Known liver abnormalities, liver cirrhosis (compensated or decompensated), known active or history of hepatitis B or C (testing not required), known gallbladder or bile duct disease, acute or chronic pancreatitis.
4. Clinical or laboratory evidence of any of the following:
5. AST/ALT > 1.5 x the upper limit of normal range (ULN), regardless of the level of total bilirubin
6. AST/ALT > 1.0 and ≤ 1.5 x ULN and total bilirubin is > ULN
7. Total bilirubin > 2 x ULN, regardless of the level of AST/ALT
8. History of photodermatitis/increased sensitivity to sun.
9. Pregnant or nursing (lactating) women.
10. Known disturbances of electrolyte balance, e.g. hypokalemia, hypocalcemia or hypomagnesemia.
11. Moderate to severe anemia (Hemoglobin level <8 g/dL).

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2019-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Novartis Investigative Site, Lambaréné, Gabon
- Ghana (2):
  - Novartis Investigative Site, Kintampo
  - Novartis Investigative Site, Navrango
- Mali (2):
  - Novartis Investigative Site, Bamako
  - Novartis Investigative Site, Sotouba
- Novartis Investigative Site, Kigali, Rwanda
- Uganda (3):
  - Novartis Investigative Site, Bushenyi
  - Novartis Investigative Site, Kampala
  - Novartis Investigative Site, Tororo

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Ndayisaba G, Yeka A, Asante KP, Grobusch MP, Karita E, Mugerwa H, Asiimwe S, Oduro A, Fofana B, Doumbia S, Jain JP, Barsainya S, Kullak-Ublick GA, Su G, Schmitt EK, Csermak K, Gandhi P, Hughes D. Hepatic safety and tolerability of cipargamin (KAE609), in adult patients with Plasmodium falciparum malaria: a randomized, phase II, controlled, dose-escalation trial in sub-Saharan Africa. Malar J. 2021 Dec 20;20(1):478. doi: 10.1186/s12936-021-04009-1. PMID 34930267
- [Derived] Schmitt EK, Ndayisaba G, Yeka A, Asante KP, Grobusch MP, Karita E, Mugerwa H, Asiimwe S, Oduro A, Fofana B, Doumbia S, Su G, Csermak Renner K, Venishetty VK, Sayyed S, Straimer J, Demin I, Barsainya S, Boulton C, Gandhi P. Efficacy of Cipargamin (KAE609) in a Randomized, Phase II Dose-Escalation Study in Adults in Sub-Saharan Africa With Uncomplicated Plasmodium falciparum Malaria. Clin Infect Dis. 2022 May 30;74(10):1831-1839. doi: 10.1093/cid/ciab716. PMID 34410358
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 10 centers in 5 countries: Mali (2), Uganda (3), Ghana (2), Gabon (1), Rwanda (2).
Pre-assignment Details: Approximately, 210 patients were planned to be randomized in six cohorts (KAE609: 150 and Coartem: 60). A total of 188 (KAE609: 137 and Coartem: 51) subjects were randomized in five cohorts. Cohort 6 was optional and never initiated. Two of the 188 randomized subjects were not treated and therefore were excluded from all analyses.
Groups:
- KAE609 10 mg SD: KAE609 10 mg once daily (QD) for 1 day
- KAE609 10 mg QD 3 Days: KAE609 10 mg (QD) for 3 days
- KAE609 25 mg SD: KAE609 25 mg once daily (QD) for 1 day
- KAE609 25 mg QD 3 Days: KAE609 25 mg once daily (QD) for 3 days
- KAE609 50 mg SD: KAE609 50 mg once daily (QD) for 1 day
- KAE609 50 mg QD 3 Days: KAE609 50 mg once daily (QD) for 3 days
- KAE609 75 mg SD: KAE609 75 mg once daily (QD) for 1 day
- KAE609 150 mg SD: KAE609 150 mg once daily (QD) for 1 day
- Pooled Coartem Control: control arm
Period: Treatment Phase
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD | Pooled Coartem Control
Started (Randomized set (RAN)) | 10 | 10 | 12 | 20 | 22 | 20 | 21 | 22 | 51
Completed | 9 | 10 | 12 | 20 | 21 | 19 | 21 | 22 | 51
Not Completed | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Technical problems | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Subject/guardian decision | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Follow-Up Phase
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD | Pooled Coartem Control
Started | 9 | 10 | 12 | 20 | 21 | 19 | 21 | 22 | 51
Completed | 9 | 10 | 12 | 20 | 21 | 19 | 20 | 22 | 50
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Subject/guardian decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized set (RAN)
Groups:
- Total: Total of all reporting groups
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD | Pooled Coartem Control | Total
Number analyzed (Participants) | 10 | 10 | 12 | 20 | 22 | 20 | 21 | 22 | 51 | 188
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.5 (10.48) | 35.4 (13.25) | 33.0 (14.96) | 31.9 (10.67) | 33.9 (12.56) | 26.4 (7.18) | 28.2 (10.25) | 30.6 (12.57) | 26.2 (9.07) | 29.7 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8 | 11 | 9 | 8 | 5 | 6 | 18 | 73
  Male | 8 | 4 | 4 | 9 | 13 | 12 | 16 | 16 | 33 | 115
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 10 | 10 | 12 | 20 | 22 | 20 | 21 | 22 | 51 | 188

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 2 CTCAE Grades Increase From Baseline in Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST)
Description: The occurrence of at least 2 CTCAE grades increase from baseline in ALT or AST during the 4 weeks study period was evaluated to characterize hepatic safety aspects of single and multiple ascending doses of KAE609 in adult malaria subjects for treatment of uncomplicated malaria caused by plasmodium falciparum. If 2 patients in a 10 patient cohort (Cohorts 1 and 2) or 3 patients in a 20 patient cohort (Cohorts 3, 4 and 5) had at least 2 CTCAE grades increase from Baseline in ALT or AST, recruitment was suspended and a review of liver safety (and any other relevant data) by safety review committee was initiated. Any further progression of the study was based on the decision by the safety review committee.
Time Frame: Day 29
Population: Safety Set (SAF). Only participants with baseline and at least one post-baseline assessment for either ALT or AST are included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD | Pooled Coartem Control
Number analyzed (Participants) | 9 | 10 | 12 | 20 | 21 | 19 | 21 | 22 | 51
Percentage of Participants | 11.1 [0.3 to 48.2] | 0 [0.0 to 30.8] | 0 [0.0 to 26.5] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 4.5 [0.1 to 22.8] | 3.9 [0.5 to 13.5]
Statistical Analysis 1: Comparison: KAE609 10 mg SD; Test type: Other; p = 0.391, Fisher Exact; 2-sided p-value results from Fisher exact test for each KAE609 treatment group compared to Pooled Coartem
Statistical Analysis 2: Comparison: KAE609 10 mg QD 3 Days; Test type: Other; p = 1, Fisher Exact; 2-sided p-value results from Fisher exact test for each KAE609 treatment group compared to Pooled Coartem
Statistical Analysis 3: Comparison: KAE609 25 mg SD; Test type: Other; p = 1, Fisher Exact; 2-sided p-value results from Fisher exact test for each KAE609 treatment group compared to Pooled Coartem
Statistical Analysis 4: Comparison: KAE609 25 mg QD 3 Days; Test type: Other; p = 1, Fisher Exact; 2-sided p-value results from Fisher exact test for each KAE609 treatment group compared to Pooled Coartem
Statistical Analysis 5: Comparison: KAE609 50 mg SD; Test type: Other; p = 1, Fisher Exact; 2-sided p-value results from Fisher exact test for each KAE609 treatment group compared to Pooled Coartem
Statistical Analysis 6: Comparison: KAE609 50 mg QD 3 Days; Test type: Other; p = 1, Fisher Exact; 2-sided p-value results from Fisher exact test for each KAE609 treatment group compared to Pooled Coartem
Statistical Analysis 7: Comparison: KAE609 75 mg SD; Test type: Other; p = 1, Fisher Exact; 2-sided p-value results from Fisher exact test for each KAE609 treatment group compared to Pooled Coartem
Statistical Analysis 8: Comparison: KAE609 150 mg SD; Test type: Other; p = 1, Fisher Exact; 2-sided p-value results from Fisher exact test for each KAE609 treatment group compared to Pooled Coartem

2. Secondary Outcome: Percentage of Participants With Polymerase Chain Reaction (PCR)-Corrected and Uncorrected Adequate Clinical and Parasitological Response (ACPR) at Day 15 and Day 29
Description: PCR-corrected and PCR-uncorrected were evaluated at Days 15 and 29 (i.e., 14 and 28 days post-dose). The presence of parasitaemia after 7 days due to reinfection was considered as PCR-corrected ACPR. Missing blood smear data at Day 15 visit and thereafter were not considered as responder for the visit unless there was a later blood smear test indicating no parasitaemia.
Time Frame: Day 15, Day 29
Population: Full Analysis Set (FAS). Only responders at each timepoint are included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD | Pooled Coartem Control
Number analyzed (Participants) | 10 | 10 | 12 | 20 | 21 | 19 | 21 | 22 | 51
Percentage of Participants
  Day 15: PCR corrected | 90.0 [55.50 to 99.75] | 90.0 [55.50 to 99.75] | 83.3 [51.59 to 97.91] | 95.0 [75.13 to 99.87] | 95.2 [76.18 to 99.88] | 84.2 [60.42 to 96.62] | 90.5 [69.62 to 98.83] | 77.3 [54.63 to 92.18] | 96.1 [86.54 to 99.52]
  Day 15: PCR uncorrected | 90.0 [55.50 to 99.75] | 90.0 [55.50 to 99.75] | 83.3 [51.59 to 97.91] | 95.0 [75.13 to 99.87] | 95.2 [76.18 to 99.88] | 84.2 [60.42 to 96.62] | 85.7 [63.66 to 96.95] | 77.3 [54.63 to 92.18] | 96.1 [86.54 to 99.52]
  Day 29: PCR corrected | 80.0 [44.39 to 97.48] | 90.0 [55.50 to 99.75] | 83.3 [51.59 to 97.91] | 90.0 [68.30 to 98.77] | 85.7 [63.66 to 96.95] | 73.7 [48.80 to 90.85] | 81.0 [58.09 to 94.55] | 68.2 [45.13 to 86.14] | 94.1 [83.76 to 98.77]
  Day 29: PCR uncorrected | 80.0 [44.39 to 97.48] | 90.0 [55.50 to 99.75] | 66.7 [34.89 to 90.08] | 80.0 [56.34 to 94.27] | 81.0 [58.09 to 94.55] | 68.4 [43.45 to 87.42] | 71.4 [47.82 to 88.72] | 59.1 [36.35 to 79.29] | 92.2 [81.12 to 97.82]

3. Secondary Outcome: Parasite Clearance Time (PCT)
Description: Parasite Clearance Time (PCT) is defined as the time from the first dose until the first total and continued disappearance of asexual parasite forms which remained at least a further 48 hours. In case a patient received rescue medication before (parasite) clearance, the time to event was censored at the first use of rescue medication.
Time Frame: Day 29
Population: Full Analysis Set (FAS). Only participants with parasite at baseline and post-baseline assessment of parasite clearance at the time point are included in the analysis.
Measure: Mean (Standard Error); unit: Hours
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD | Pooled Coartem Control
Number analyzed (Participants) | 10 | 10 | 12 | 20 | 21 | 19 | 21 | 22 | 51
Hours | 26.8 (5.44) | 27.7 (4.96) | 14.0 (2.63) | 11.4 (1.82) | 11.1 (1.58) | 9.8 (0.97) | 8.7 (0.97) | 8.0 (1.09) | 36.2 (3.72)

4. Secondary Outcome: Fever Clearance Time (FCT)
Description: Fever Clearance Time (FCT) is defined as the time from the first dose until the first time the axillary body temperature decreased below and remained below 37.5°C axillary or 38.0°C oral/tympanic/rectal for at least a further 24 hours. In case a patient received rescue medication before (fever) clearance, the time to event was censored at the first use of rescue medication.
Time Frame: Day 29
Population: Full Analysis Set (FAS). Only participants with fever at baseline and post-baseline assessment of fever clearance at the time point are included in the analysis.
Measure: Mean (Standard Error); unit: Hours
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD | Pooled Coartem Control
Number analyzed (Participants) | 10 | 10 | 12 | 20 | 21 | 19 | 21 | 22 | 51
Hours | 3.9 (NA) — NA: Not Estimable due to number of events censored | 2.0 (0.02) | NA (NA) — NA: Not Estimable due to number of events censored | 22.0 (14.03) | 2.4 (0.93) | 7.2 (1.47) | 5.7 (2.02) | 9.9 (3.88) | 13.0 (4.29)

5. Secondary Outcome: Time to Recrudescence and Reinfection at Study Day 29
Description: Time to recrudescence is calculated from the date of first study medication to the date of first event. Participants without recrudescence/reinfection after Day 7 are censored at the time of treatment failure or at the time of last parasite assessment if no treatment failure occured.
Time Frame: Day 29
Population: Full Analysis Set (FAS). Only participants with clearance of initial infection before Day 15 and recrudescence/reinfection are included in the analysis.
Measure: Number (95% Confidence Interval); unit: Event probability
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD | Pooled Coartem Control
Number analyzed (Participants) | 8 | 10 | 12 | 20 | 21 | 19 | 21 | 22 | 51
Event probability
  Recrudescence: number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 5 | 3 | 7 | 1
  Recrudescence | 12.5 [1.86 to 61.30] | 10.0 [1.47 to 52.70] | 16.7 [4.45 to 51.83] | 10.0 [2.60 to 34.40] | 16.0 [5.42 to 41.93] | 26.3 [11.90 to 52.11] | 15.9 [5.40 to 41.67] | 32.5 [16.93 to 56.43] | 2.4 [0.34 to 15.72]
  Reinfection: number analyzed (Participants) | 0 | 0 | 2 | 2 | 1 | 1 | 2 | 2 | 1
  Reinfection |  |  | 25.0 [6.91 to 68.52] | 14.3 [3.78 to 46.06] | 5.0 [0.72 to 30.53] | 10.0 [1.47 to 52.70] | 10.3 [2.67 to 35.25] | 13.3 [3.51 to 43.61] | 2.4 [0.34 to 15.72]

6. Secondary Outcome: Maximum Peak Observed Concentration (Cmax)
Description: Maximum Peak Observed Concentration (Cmax)
Time Frame: Day 1, Day 3
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD
Number analyzed (Participants) | 9 | 10 | 12 | 20 | 21 | 19 | 20 | 22
ng/mL
  Day 1 | 179 (38.2) | 185 (51.2) | 379 (42.1) | 503 (44.3) | 773 (32.4) | 828 (35.4) | 1270 (41.3) | 2360 (28.5)
  Day 3: number analyzed (Participants) | 0 | 10 | 0 | 20 | 0 | 19 | 0 | 0
  Day 3 |  | 235 (37.0) |  | 655 (27.9) |  | 1210 (30.7) |  |

7. Secondary Outcome: Tmax
Description: Tmax
Time Frame: Day 1, Day 3
Population: PK Analysis Set
Measure: Median (Full Range); unit: Hour
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD
Number analyzed (Participants) | 9 | 10 | 12 | 20 | 21 | 19 | 20 | 22
Hour
  Day 1 | 4.00 [1.02 to 12.10] | 3.92 [1.03 to 6.17] | 4.01 [2.00 to 8.33] | 4.25 [2.00 to 23.80] | 4.12 [1.97 to 10.00] | 4.12 [2.00 to 6.13] | 6.01 [3.97 to 12.30] | 8.07 [1.00 to 24.10]
  Day 3: number analyzed (Participants) | 0 | 10 | 0 | 20 | 0 | 19 | 0 | 0
  Day 3 |  | 52.7 [50.00 to 60.60] |  | 52.1 [49.90 to 59.60] |  | 52.0 [50.00 to 60.50] |  |

8. Secondary Outcome: AUC0-24
Description: AUC0-24
Time Frame: Day 1, Day 3
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD
Number analyzed (Participants) | 9 | 10 | 12 | 20 | 21 | 19 | 20 | 22
h*ug/mL
  Day 1: number analyzed (Participants) | 9 | 9 | 12 | 16 | 21 | 14 | 20 | 22
  Day 1 | 2.77 (48.9) | 2.59 (38.0) | 5.14 (52.5) | 8.39 (45.1) | 11.6 (37.7) | 15.6 (27.2) | 21.4 (41.5) | 40.4 (26.6)
  Day 3: number analyzed (Participants) | 0 | 10 | 0 | 20 | 0 | 19 | 0 | 0
  Day 3 |  | 3.90 (38.5) |  | 10.9 (29.7) |  | 21.6 (31.3) |  |

9. Secondary Outcome: Half-life (T^1/2)
Description: Half-life (T^1/2)
Time Frame: Upto day 15 post dose
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | KAE609 10 mg SD | KAE609 10 mg QD 3 Days | KAE609 25 mg SD | KAE609 25 mg QD 3 Days | KAE609 50 mg SD | KAE609 50 mg QD 3 Days | KAE609 75 mg SD | KAE609 150 mg SD
Number analyzed (Participants) | 9 | 10 | 12 | 20 | 21 | 19 | 20 | 22
Hour
  Day 1: number analyzed (Participants) | 8 | 3 | 11 | 2 | 20 | 2 | 17 | 21
  Day 1 | 24.4 (8.70) | 18.5 (6.24) | 35.1 (13.9) | 17.4 (3.27) | 31.5 (17.4) | 32.8 (5.05) | 25.3 (8.94) | 29.9 (12.5)
  Day 3: number analyzed (Participants) | 0 | 8 | 0 | 18 | 0 | 17 | 0 | 0
  Day 3 |  | 32.4 (14.8) |  | 30.1 (14.0) |  | 29.9 (22.0) |  |

ADVERSE EVENTS:
Time Frame: All AEs reported in this record are treatment emergent AEs, collected from date of First Patient First Treatment until the completion of the safety follow-up ( 30 days after the Last Patient Last Treatment ) up to approximately 2 years.
Groups:
- KAE609 10mg SD: KAE609 10mg SD
- KAE609 10mg QD@3 Days: KAE609 10mg QD@3 days
- KAE609 25mg SD: KAE609 25mg SD
- KAE609 25mg QD@3 Days: KAE609 25mg QD@3 days
- KAE609 50mg SD: KAE609 50mg SD
- KAE609 50mg QD@3 Days: KAE609 50mg QD@3 days
- KAE609 75mg SD: KAE609 75mg SD
- KAE609 150mg SD: KAE609 150mg SD
- Pooled Coartem: Pooled Coartem
Arm/Group | KAE609 10mg SD | KAE609 10mg QD@3 Days | KAE609 25mg SD | KAE609 25mg QD@3 Days | KAE609 50mg SD | KAE609 50mg QD@3 Days | KAE609 75mg SD | KAE609 150mg SD | Pooled Coartem
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/12 | 0/20 | 0/21 | 0/19 | 0/21 | 0/22 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/12 | 0/20 | 0/21 | 1/19 | 2/21 | 1/22 | 1/51
Other Adverse Events (participants affected / at risk) | 9/10 | 8/10 | 10/12 | 10/20 | 9/21 | 16/19 | 15/21 | 12/22 | 25/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KAE609 10mg SD (N=10) | KAE609 10mg QD@3 Days (N=10) | KAE609 25mg SD (N=12) | KAE609 25mg QD@3 Days (N=20) | KAE609 50mg SD (N=21) | KAE609 50mg QD@3 Days (N=19) | KAE609 75mg SD (N=21) | KAE609 150mg SD (N=22) | Pooled Coartem (N=51)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KAE609 10mg SD (N=10) | KAE609 10mg QD@3 Days (N=10) | KAE609 25mg SD (N=12) | KAE609 25mg QD@3 Days (N=20) | KAE609 50mg SD (N=21) | KAE609 50mg QD@3 Days (N=19) | KAE609 75mg SD (N=21) | KAE609 150mg SD (N=22) | Pooled Coartem (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Treatment failure (General disorders) | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 2
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 3 | 2
Malaria (Infections and infestations) | 1 | 0 | 2 | 4 | 4 | 5 | 5 | 9 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parasitic gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 5 | 1 | 1 | 2 | 2 | 5 | 0 | 9
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03334747/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT03334747/SAP_001.pdf